CLINICAL TRIAL: NCT01435590
Title: Endocervical Evaluation With the Curette Versus Cytobrush for the Diagnosis of Dysplasia of the Uterine Cervix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Manuela Undurraga Malinverno, Medecin Interne, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CER 11-029
Record Dates: First submitted 2011-09-13; First posted 2011-09-16 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Cervical Dysplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Curette v/s endocervical brush

SUMMARY:
OBJECTIVE: to compare endocervical brushing with endocervical curettage with respect to diagnostic and patient discomfort.

METHOD: women referred to colposcopy because of abnormal Papanicolaou tests will be randomized to endocervical sampling with either a metal curette (endocervical curettage -ECC) or and endocervical brush. All samples will be submitted for histological study.

ELIGIBILITY:
Inclusion Criteria:

* French-speaking
* 21 years or older
* Attending our colposcopy clinic
* Need for endocervical evaluation
* Full autonomy or capacity to understand the procedures

Exclusion Criteria:

* Pregnancy
* Absence of uterus
* History of DES exposure in utero

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Specimen adequacy | 09/2011 - 05/2012 (1 year)
  Cytological and histological interpretation of the endocervical brush specimens will then be performed, while for the endocervical currete specimens only histological interpretation will be done. The adequacy of the specimens will be based on the quantity of endocervical cells present (< or ≥ 20 endocervical cells), the quantity of histological material (< or ≥ 3 epithelial stripes) and the quality of histological material (absence or presence of lamina propia).

SECONDARY OUTCOMES:
Patient discomfort | 09/2011 to 05/2012 (8 months)
  To evaluate the degree of patient discomfort, patients will be requested to complete a questionnaire once the exam has been completed. The main acceptance variables will be degree of helplessness, pain (on visual analog scales), willingness to undergo the test again, and overall satisfaction. Once the exam has been completed, the doctor performing the sampling will answer a questionnaire indicating his/her perception of the exam (patient's pain, technical difficulty performing the exam, doctors acceptability of the exam).

REFERENCES:
- [Derived] Undurraga M, Catarino R, Navarria I, Ibrahim Y, Puget E, Royannez Drevard I, Pache JC, Tille JC, Petignat P. User perception of endocervical sampling: A randomized comparison of endocervical evaluation with the curette vs cytobrush. PLoS One. 2017 Nov 6;12(11):e0186812. doi: 10.1371/journal.pone.0186812. eCollection 2017. PMID 29107949